CLINICAL TRIAL: NCT06664255
Title: High Prevalence of Secondary Arterial Hypertension (HIPRESH) with Prospective Systematic Screening
Brief Title: High Prevalence of Secondary Arterial Hypertension (HIPRESH) with Prospective Systematic Screening in a Cohort of Consecutive Hypertensive Patients Referring to Regional Specialized Center
Acronym: HIPRESH
Status: Completed | Type: Observational
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Gian Paolo Rossi, MD, FAHA, FACC, Principal Investigator, University Hospital Padova
Other Study IDs: F 004
Record Dates: First submitted 2024-10-22; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hypertension; Hypertension Resistant to Conventional Therapy; Secondary Hypertension to Endocrine Disorders; Secondary Hypertension; Secondary Hypertension Renal Arterial
Keywords: Secondary Hypertension; Primary Aldosteronism; Causes; Hyperaldosteronism; Hypertension, Renovascular; Hypertension, Renal; Essential Hypertension; Prevalence
MeSH Terms: conditions — Hypertension; Hypertension Resistant to Conventional Therapy; Hyperaldosteronism; Hypertension, Renovascular; Hypertension, Renal; Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood serum samples and 24h urine samples will be obtained by all patients. Further examination will be obtained as required by the diagnostic workup.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hypertensive patients: Consecutive hypertensive patients referring to our center, and undergoing systematic diagnostic workup for secondary causes of hypertension

SUMMARY:
Hypertensive Patients referring to our center will undergo a systematic diagnostic workup aimed at finding the cause(s) of their high blood pressure. Information prospective and retrospectively obtained will be analyzed while guaranteeing anonymity.

DETAILED DESCRIPTION:
The Investigators will retrospectively enroll consecutive patients attending the outpatient clinic of the Specialized Hypertension Center at the Department of Medicine of the University of Padua from January 1 st 2017 to January 31 st 2023. The data obtained from the review of clinical chart and findings from biochemical and radiological examinations will be recorded in a secured database and will be analyzed in an anonymized and aggregated form.

Per Investigators' practice, during the first visit, patients attending our Referral Center undergo a complete clinical evaluation entailing extensive medical history and supine and standing office blood pressure measurement, ECG and are offered a screening for secondary hypertension. To this end, patients are usually switched to treatment with a long-acting calcium-channel blocker, mostly verapamil slow-release and/or doxazosin, for at least 6 weeks beforebiochemical testing.

From 2020, based on the results of the "Effects of Mineralocorticoid and AT1 Receptor Antagonism on the Aldosterone-Renin Ratio in Primary Aldosteronism" (EMIRA), 13 those with difficult-to-control hypertension and/or hypokalemia also received a mineralocorticoid receptor antagonist (MRA). As per institutional rules, at the Investigators' University Hospital all the patients are requested to sign a written consent for the processing of their data in an anonymized way for educational and research purpose. All the patients will receive exhaustive information about the need of screening for secondary hypertension, which entailed good clinical practice.

Biochemical data that will be recorded include serum Na + , K + , and ionized Ca 2+ levels, plasma active renin concentration (DRC), aldosterone concentration (PAC), used to compute the aldosterone-renin ratio (ARR), 24h urine Na + , K + , and Ca 2+ excretion, metanephrine and normetanephrine excretion in acidified urines, serum parathyroid hormone, thyroid-stimulating hormone, and free triiodothyronine and free thyroxine. The Investigators will also record data from renal Doppler ultrasonography, sleep questionnaires for sleep apnoea, sleep fragmentation, and daytime sleepiness, when performed. In patients who underwent second level imaging tests, e.g. abdomen MRI, CT or angio-CT and subtyping by adrenal vein sampling (AVS) or full poly-somnography, data from these additional tests will be registered.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 and >/= 85 years

Exclusion Criteria:

* absence of a complete diagnostic work-up due to poor overall clinical conditions or lack of a clear benefit from it
* unwillingness or failure to complete the full diagnostic work-up and/or to attend the outpatient clinic follow-up visits after the first evaluation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients refering to our center
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Patients with a Diagnosis of Secondary hypertension | From enrolment to assessment of cure/target treatment at follow up, an average of 1 year.
  Conclusive diagnosis of secondary hypertension based on the availble gold standard confirmed by assessment of cure/improvement after target treatment at follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Rossi, MD, Principal Investigator — University of Padova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azizi M, Sapoval M, Gosse P, Monge M, Bobrie G, Delsart P, Midulla M, Mounier-Vehier C, Courand PY, Lantelme P, Denolle T, Dourmap-Collas C, Trillaud H, Pereira H, Plouin PF, Chatellier G; Renal Denervation for Hypertension (DENERHTN) investigators. Optimum and stepped care standardised antihypertensive treatment with or without renal denervation for resistant hypertension (DENERHTN): a multicentre, open-label, randomised controlled trial. Lancet. 2015 May 16;385(9981):1957-65. doi: 10.1016/S0140-6736(14)61942-5. Epub 2015 Jan 26. PMID 25631070
- [Background] Rossi GP, Bagordo D, Rossi FB, Pintus G, Rossitto G, Seccia TM. 'Essential' arterial hypertension: time for a paradigm change. J Hypertens. 2024 Aug 1;42(8):1298-1304. doi: 10.1097/HJH.0000000000003767. Epub 2024 May 8. PMID 38748508